CLINICAL TRIAL: NCT05527405
Title: Efficacy of Caregiver Training Program in Enhancing Caregiver and Patient Outcomes in Visual Mapping Assistive Technology
Brief Title: Efficacy of Caregiver Training Program in Enhancing Caregiver and Patient Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MapHabit, Inc. (Industry)
Responsible Party: Principal Investigator, Stuart Zola, Chief Scientific Officer, MapHabit, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Fast Track - CTP (NIH-SBIR)
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease; Dementia; Caregiver Burden; Assistive Technology
Keywords: Alzheimer Disease; Dementia; Caregiver Burden; Activities of Daily Living; Assistive Technology
MeSH Terms: conditions — Alzheimer Disease; Dementia; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: The study will be a randomized controlled clinical trial in which two conditions will be investigated: a control and an experimental condition.
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistical analyses of all data will be carried out independently of investigators by a biostatistical resource department of an academic health center for validation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caregiver Training Program (Experimental): This condition will involve the implementation of an assistive technology software (named the MapHabit System) with an added Caregiver Training Program into the daily care of individuals with mild to moderate stages of Alzheimer's disease and related dementias. The MapHabit System (MHS) is a commercially available visual mapping software application that utilizes visual, audio, and text media to create step-by-step visual guides to assist individuals and their caregivers in structuring and accomplishing activities of daily living (ADLs). The application will be made available to families through compatible tablets.
  Interventions: Device: The MapHabit System
- The MapHabit System (Active Comparator): This control condition will act as the active comparator to the experimental condition. The same assistive technology, the MapHabit System, will be given to a separate group of participants. The difference here will be that the software will be a version that does not include the caregiver training program.
  Interventions: Device: The MapHabit System

INTERVENTIONS:
Device: The MapHabit System — The MapHabit System (MHS) is a commercially available visual mapping software application that utilizes visual, audio, and text media to create step-by-step visual guides to assist individuals and their caregivers in structuring and accomplishing activities of daily living (ADLs). The goal of the application is to develop and facilitate habits and routines using structured visual and auditory stimuli that can be customized by the user and can include educational and lesson-based material in addition to ADLs. The application will be made available through tablets. Depending on the condition, participants will receive a specific version of the application. The experimental condition will receive the version that incorporates gamified structure and the Caregiver Training Program.
  The MHS is a general wellness product. This functionality is not a regulated medical device.

SUMMARY:
As part of Phase II of the NIH SBIR grant, the study will conduct a randomized controlled clinical trial in which the MapHabit system (MHS) will offer a caregiver training product that is linked to MHS, an Alzheimer's disease or related dementias (AD/ADRD) assistive technology product that uses visual maps to improve a patient's behavior and sense of autonomy. MapHabit's combined areas of focus, i.e., offer a single integrated product to address the caregiver and the person under this caregiver's care, are unique and will create a new standard in the field to reduce caregiver burden in the setting of caring for individuals with AD/ADRD. Additionally, the study will integrate enhanced user support modules, i.e., gamifying, dashboarding, and social networking, to improve the Caregiver Training Program (CTP) experience.The study will be a randomized controlled clinical trial, in which two conditions will be investigated: 1) control condition in which the MHS alone is incorporated in the participant's daily care and 2) experimental condition in which the MHS+CTP is implemented into the daily care received by participants. The sample size will be a total of 50 patient-caregiver dyads, 25 in each condition. The study duration will be a 6-month intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individual diagnosed with Alzheimer's disease or other related dementia (ADRD) in their mild to moderate stage of impairment
* Participating caregiver of individual with dementia must be the primary caregiver
* Proficient in English

Exclusion Criteria:

* Individual not diagnosed with ADRD
* Participating caregiver of individual with dementia is NOT the primary caregiver
* Not proficient in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-24 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in User Interaction and Engagement from baseline at 6 months | Pre-Post: The instrument will be administered to the participants at baseline, post-intervention (6 months)
  18-item quality-of-life questionnaire (QoL-18) evaluates a range of participants' behaviors, including mood, engagement, and memory at the end of the study compared to before the use of the MHS. The instrument is scored on a Likert Scale, ranging from 1-10. A higher number indicates better outcome.
Change in Zarit Burden Assessment Caregiver Strain instrument from baseline at 6 months | Pre-Post: The instrument will be administered to the participants at baseline, post-intervention (6 months)
  18-item questionnaire assessing the various stresses caregivers experienced relating to caring for an individual with cognitive impairment. The total score ranges from 0-72, with a higher score reflecting higher stress and burden on the caregiver.
Change in Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL) from baseline at 6 months | Pre-Post: The instrument will be administered to the participants at baseline, post-intervention (6 months)
  Assesses an individual with dementia's ability to carry out activities of daily living. The total score ranges from 0-53, with a higher score representing better performance in completing activities of daily living by the individual with dementia.
Change in Quality of Life - 18 (QoL-18) from baseline at 6 months | Pre-Post: The instrument will be administered to the participants at baseline, post-intervention (6 months)
  18-item quality-of-life questionnaire (QoL-18) evaluated a range of participants' behaviors, including mood, engagement, and memory at the middle and end of the study compared to before the use of the MHS. The instrument is scored on a Likert Scale, ranging from 1-10. A higher number indicates better outcome.
Change in Brief Quality of Life - 8 (QoL-8) from baseline at 6 months | Pre-Post: The instrument will be administered to the participants at baseline, post-intervention (6 months)
  8-items selected from the Wisconsin Quality of Life Caregiver Questionnaire evaluated a range of participants' behaviors, including mood, engagement, and memory at the middle and end of the study compared to before the use of the MHS. The instrument is scored on a Likert Scale, ranging from 1-10. A higher number indicates better outcome.
Change in Caregiver Self-Assessment Questionnaire from baseline at 6 months | Pre-Post: The instrument will be administered to the participants at baseline, post-intervention (6 months)
  12-item, caregiver self-report measure of stress levels

SECONDARY OUTCOMES:
2-item Satisfaction Scale (SS-2) | The instrument was administered to the participants after the completion of the study duration (i.e., assessed at 6 months)
  Quantifies caregivers' endorsements to two survey questions: How satisfied were they with the MHS? Would they recommend MHS to others? Both questions are scored on a 10-point scale, with a higher value reflecting a better outcome/experience.
Pain and Sleep Questionnaire | Pre-Post: The assessment will be administered at baseline, post-intervention (6 months)
  5-item questionnaire developed to assess the impact of pain on quality of sleep
Generalized Anxiety Disorder (GAD7) Scale | Pre-Post: The assessment will be administered at baseline, post-intervention (6 months)
  7-item questionnaire used as an initial screening tool for generalized anxiety disorder
Anger Management Scale | Pre-Post: The assessment will be administered at baseline, post-intervention (6 months)
  12-item questionnaire designed to monitor and evaluate progress in controlling and managing anger

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Zola, Principal Investigator — MapHabit, Inc.
Locations (1):
- MapHabit, Inc., Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to szola@maphabit.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Boatman F, Golden M, Jin J, Kim Y, Law S, Lu A, Merriam N, Zola S. Assistive technology: Visual mapping combined with mobile software can enhance quality of life and ability to carry out activities of daily living in individuals with impaired memory. Technol Health Care. 2020;28(2):121-128. doi: 10.3233/THC-191980. PMID 31796718
- [Background] Kelleher J, Zola S, Cui X, Chen S, Gerber C, Parker MW, Davis C, Law S, Golden M, Vaughan CP. Personalized Visual Mapping Assistive Technology to Improve Functional Ability in Persons With Dementia: Feasibility Cohort Study. JMIR Aging. 2021 Oct 19;4(4):e28165. doi: 10.2196/28165. PMID 34269690
- [Background] Parker MW, Davis C, White K, Johnson D, Golden M, Zola S. Reduced care burden and improved quality of life in African American family caregivers: Positive impact of personalized assistive technology. Technol Health Care. 2022;30(2):379-387. doi: 10.3233/THC-213049. PMID 34334439